CLINICAL TRIAL: NCT01158300
Title: Phase I and Pharmacokinetic Trial of PTC299 in Pediatric Patients With Refractory or Recurrent CNS Tumors
Brief Title: PTC299 in Treating Young Patients With Refractory or Recurrent Primary Central Nervous System Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000680634; U01CA081457 (NIH); PBTC-031 (Other: Pediatric Brain Tumor Consortium); PTC299-ONC-010-PBT (Other: PTC Therapeutics)
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent childhood malignant germ cell tumor; recurrent childhood brain stem glioma; recurrent childhood brain tumor; recurrent childhood central nervous system embryonal tumor; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood ependymoma; recurrent childhood medulloblastoma; recurrent childhood pineoblastoma; recurrent childhood rhabdomyosarcoma; recurrent childhood spinal cord neoplasm; recurrent childhood subependymal giant cell astrocytoma; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood visual pathway glioma; childhood central nervous system choriocarcinoma; childhood central nervous system germ cell tumor; childhood central nervous system germinoma; childhood central nervous system mixed germ cell tumor; childhood central nervous system teratoma; childhood central nervous system yolk sac tumor; childhood astrocytoma; childhood medulloepithelioma; childhood meningioma; childhood mixed glioma; childhood oligodendroglioma; childhood pineal parenchymal tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Familial ependymoma; Medulloblastoma; Spinal Cord Neoplasms; Optic Nerve Glioma; Meningioma; Oligodendroglioma | interventions — emvododstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: VEGF inhibitor PTC299 — This is a dose escalation study. Study participants will receive .6 or 1.2 mg/kg orally twice daily or 1.2, 1.5, or 2.0 mg/kg orally three times daily for four consecutive weeks (a course). In the absence of unacceptable toxicity or disease progression, treatment may continue for up to 12 courses (approximately one year)

SUMMARY:
RATIONALE: PTC299 may stop the growth of tumor cells by blocking blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and the best dose of PTC299 in treating young patients with recurrent or refractory primary central nervous system tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the maximum-tolerated dose and the recommended phase II dose of VEGF inhibitor PTC299 (PTC299) in pediatric patients with recurrent or progressive primary central nervous system (CNS) tumors.
* To evaluate and characterize the adverse events associated with this regimen in these patients.
* To evaluate and characterize the pharmacokinetics and pharmacodynamics of this regimen in these patients.

Secondary

* To investigate the relationships between PTC299 plasma exposure and other outcomes measures.
* To evaluate the antitumor activity of this regimen in these patients.
* To evaluate changes in angiogenic and inflammatory markers in the blood and the relationship between these changes and other outcome measures.
* To obtain preliminary evidence of biologic activity of PTC299 by using magnetic resonance diffusion to assess tumor cellularity.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive oral VEGF inhibitor PTC299 twice or thrice daily. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and periodically during study for pharmacokinetic and pharmacodynamic studies by ELISA.

After completion of study therapy, patients are followed up for 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of primary central nervous system (CNS) malignancy at time of diagnosis or recurrence

  * Histology verification not required for intrinsic brain stem tumors and optic pathway gliomas

    * Must have radiographic evidence of progression
* Recurrent, progressive, or refractory disease to standard therapy and for which there is no known curative therapy

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% (patients > 16 years of age) OR Lansky PS 50-100% (patients ≤ 16 years of age)
* Body weight ≥ 15 kg and ≤ 100 kg
* Patients with neurological deficits allowed provided they are stable for ≥ 1 week
* Able to swallow capsules
* ANC ≥ 1,000/μL (unsupported)
* Platelet count ≥ 100,000/μL (unsupported)
* Hemoglobin ≥ 8 g/dL (may be supported)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70 mL/min/1.73 m^2 OR serum creatinine normal based on age as follows:

  * 0.8 mg/dL (≤ 5 years of age)
  * 1.0 mg/dL (> 5 to ≤ 10 years of age)
  * 1.2 mg/dL (> 10 to ≤ 15 years of age)
  * 1.5 mg/dL (> 15 years of age)
* Urine protein/creatinine ratio < 1.0
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN
* Albumin ≥ 2.5 g/dL
* PT and activated PTT ≤ 1.2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No clinically significant unrelated systemic illness that would compromise the patient's ability to tolerate protocol therapy, or would likely interfere with the study procedures or results, including any of the following:

  * Serious infections including ongoing systemic bacterial, fungal, or viral infection
  * Significant cardiac, pulmonary, hepatic, or other organ dysfunction
* Willing and able to comply with schedule visits, drug administration plan, laboratory tests, including pharmacokinetic and pharmacodynamic assessments, or other study procedures
* No known coagulopathy or bleeding diathesis
* No known history of drug-induced liver injury
* No CNS, pulmonary, gastrointestinal, or urinary bleeding within the past month
* No uncontrolled systemic hypertension (systolic BP or diastolic BP > 95% percentile for age)
* No alcohol or drug addiction
* Able to tolerate periodic MRI scans and gadolinium contrast

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from the acute toxic of all prior therapy (excluding alopecia and neurotoxicity)
* At least 3 weeks since prior myelosuppressive anticancer chemotherapy (6 weeks for nitrosourea)
* At least 14 days since prior investigational or biological agent

  * At least 3 half-lives since prior biological agents that have a prolonged half-life
* At least 3 half-lives since prior monoclonal antibody
* At least 2 weeks since prior local palliative radiotherapy
* At least 6 weeks since prior total-body irradiation, craniospinal radiotherapy, or radiotherapy to ≥ 50% of the pelvis
* At least 90 days since prior allogeneic bone marrow transplantation

  * No active graft-versus-host disease
* Concurrent dexamethasone or other corticosteroids allowed provided dose is stable for ≥ 7 days
* At least 1 week since prior colony-forming growth factors (e.g., filgrastim, sargramostim, erythropoietin)

  * At least 14 days since long-acting colony-forming growth factor formulations (e.g., pegfilgrastim)
* More than 4 weeks since prior major surgical procedures

  * More than 2 weeks since prior intermediate surgical procedures
  * More than 7 days since minor surgical procedures
* No other concurrent anticancer or investigational drug therapy

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2010-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose | First four weeks of treatment
Adverse events | From the first day of treatment until 30 days after the last dose

SECONDARY OUTCOMES:
Percentage of study participants with complete response or partial response to the study treatment | Every 8 weeks
  Brain images to assess partial or complete response are performed every 8 weeks after the first dose of the study drug.
Pharmacokinetics | Day 1 and day 28 of course 1
  Blood samples from study participants will be collected on day 1 and day 28 of course 1 for standard full pharmacokinetic studies.
Change from baseline in blood angiogenic markers and cytokines at discontinuation or completion of treatment | Before the first dose of drug on day 1 of course 1 and at the discontinuation or completion of treatment
  Blood samples will be collected and analyzed on Day 1 of pre-AM dosing at baseline and at the discontinuation or completion of treatment. Changes from baseline in blood angiogenic markers and cytokines (VEGF-A, VEGF-C, VEGF-D, PlGF, VEGFR-1, VEGFR-2, IL-6, and IL-8) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Roger J. Packer, MD, Principal Investigator — Children's National Research Institute
Locations (8):
- United States (8):
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas